CLINICAL TRIAL: NCT04121832
Title: Biofeedback Training, Efficacy Evaluation of Fibromyalgia Treatment, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Mauro Giovanni Carta, Principal Investigator, University of Cagliari
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PG/2019/6248
Record Dates: First submitted 2019-06-06; First posted 2019-10-10 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Biofeedback, Psychology
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a controlled clinical trial with crossover and comparison between usual care and biofeedback training, plus usual care
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Case (Experimental): 32 women with fibromyalgia diagnosis corresponding to the diagnostic criteria of the American College of Rheumatology (ACR) will be taken in charge at the pain therapy centre of San Giovanni di Dio Hospital. All patients over the age of 18 will be included.
  Other patients with rheumatologic diagnoses in comorbidity with fibromyalgia will be considered exclusion criteria/will be excluded. Patients with cognitive difficulties and / or diagnoses of intellectual disability and male patients will not be included in the study. In addiction to standard therapies, the sample will be treated with 10 sessions of biofeedback training.
  Interventions: Device: Biofeedback training treatment in Fibromyalgia, a pilot study
- Controls (Active Comparator): 32 women with fibromyalgia diagnosis corresponding to the diagnostic criteria of the American College of Rheumatology (ACR) will be taken in charge at the pain therapy centre of San Giovanni di Dio. All patients over the age of 18 will be included. Other patients with rheumatologic diagnoses in comorbidity with fibromyalgia will be considered exclusion criteria/will be excluded. Moreover, patients with cognitive difficulties and / or diagnoses of mental retardation and male patients will not be included in the study. The sample will be treated only with standard therapies without the use of biofeedback training
  Interventions: Other: Control (treatment as usual)

INTERVENTIONS:
Device: Biofeedback training treatment in Fibromyalgia, a pilot study — The selected sample will undergo 10 total Biofeedback Training sessions, once a week. Each session will last 45 minutes. The total duration of the treatment will be 10 weeks
  Arms: Case
Other: Control (treatment as usual) — The sample will be treated only with standard therapies without the use of biofeedback training for 10 weeks
  Arms: Controls

SUMMARY:
Biofeedback equipment is classified by the Food and Drug Administration (FDA) as medical device class II and this type of equipment/treatment has shown evidence regarding stress management.

In fibromyalgia. The main objective of the study is to verify the feasibility of an HVR biofeedback training protocol in patients with fibromyalgia, and also to verify improvement induced by the technique in relation to: Quality of life; Quality of sleep; Perception of pain; Depressive symptomatology; Anxious symptomatology.

DETAILED DESCRIPTION:
Background and rationale of study

Fibromyalgia (FM) is a chronic disease, it is characterised by persistent and diffused musculoskeletal pain with not well defined etiology. Fibromyalgia often occurs in comorbidity with other functional, organic and psychiatric pathologies. The main clinical manifestation of FM is pain, which is predominantly described by people with fibromyalgia as a burning sensation, stiffness, contracture and tension. Pain varies depending on moments of the day, activity levels, weather conditions, sleep cycle and perceived distress. Patients suffering from fibromyalgia commonly have functional disorders, including persistent fatigue,dysregulated sleep, cognitive slowness, bowel disorders, paresthesia. Futhermore, fibromyalgia occurs in comorbidity with depression with a percentage that varies between 22% and 80% (3,4). Moreover, some patients with fibromyalgia have anxiety disorder and other syndromes related to stress as irritable bowel. The prevalence of fibromyalgia in general population is 2%, with a peak of onset between 45-60 years. The gender prevalence varies between 0.5% and 5%, it is more common between women (~ 4.2%) than men (~0.2%).

Fibromyalgia has an important impact on the quality of life. Biofeedback is one of the medical devices used for the treatment of fibromyalgia, that aimes to riduce the typical symptoms and improve QoL.

Biofeedback allows to learn self-regulation of some physiological processes through feedback of recorded parameters and the goal is improving health and its performances.

Biofeedback measures muscle activity, skin temperature, electrodermal activity (sudoriparous glands activity), respiration, heart rate, blood pressure, electrical brain activity and bloodstream, it also gives a quick feedback of those personal measurements to the patient, in this way biofeedback teaches people to have a more active role in maintaining a good personal, mental and physical health (quickly and thoroughly it give person feedback of activity and biofeedback teaches people to take a more active role in maintaining personal health and mental health and physical health).

Biofeedback equipment is classified by the Food and Drug Administration (FDA) as medical device class II and this type of equipment/treatment has shown evidence regarding stress management (evidence were shown as regards stress menagement).

In fibromyalgia, the greatest benefits from using biofeedback are: improvement of sleep quality, improvement of self- efficacy, improvement of pain threshold, and improvement of emotional adjustment. In particular, a study conducted with HRV biofeedback, in which the sample learned resonance frequency breathing, showed dicreases in depression and pain and improved the person's system functioning.

Study objectives

The main objective of the study is to verify the feasibility of an HVR biofeedback training protocol in patients with fibromyalgia, and also to produce a preliminary measurement of the possible improvement induced by the technique in relation to:Quality of life; Quality of sleep; Perception of pain; Depressive symptomatology; Anxious symptomatology This measure will be useful to estimate the expected improvement in future case-control studies. Study design

This is a controlled clinical trial with crossover and comparison between usual care and biofeedback training, plus usual care.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with fibromyalgia afferent to the clinic of pain therapy of San Giovanni hospital in Cagliari, Sardegna. Psychiatric comorbidities have no exclusion criterion

Exclusion Criteria:

- Patients with cognitive difficulties and/or diagnoses of mental retardation and male patients will not be included in the study. Male patients will be excluded because the diagnosy of FM is infrequent in male patients and it was decided not to have bias because of the low amount of patients included in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Quality of sleep, Sleep scale from the medical study (MOS),change is being assessed | T0 (0 weeks); T1 (10 weeks); T2 (22 weeks); T3 (34 weeks)
  Self-assessment questionnaire consisting of 12 items and is aimed at evaluating certain fundamental parameters in sleep disorders such as sleep, sleep continuity, sleep duration, sleepiness and breathing disorders during sleep. The total score is on the scale ranges from 0 to 100. Higher scores indicate more disturbed sleep
Fibromyalgia Impact Questionnaire (FIQ), change is being assessed | T0 (0 weeks); T1 (10 weeks); T2 (22 weeks); T3 (34 weeks)
  self-administered questionnaire, consisting of 20 questions, divided into three parts: ability to carry out activities of daily life; number of days in the last week in which the patient has felt good and in which he has not been able to carry out his work due to the symptoms of FM. Questions 4 to 10 relate to the extent of FM interference with one's work, the intensity of pain and fatigue, the quality of the night's rest, the intensity of stiffness and the presence of anxiety or depression; responses range from 0 (no disturbance) to 10 (very important disorder), marked on a horizontal linear scale. The maximum FIQ score, corresponding to the highest degree of disability, is 100
Patient Health Questionnaire-9 (PHQ-9), change is being assessed | T0 (0 weeks); T1 (10 weeks); T2 (22 weeks); T3 (34 weeks)
  Short self-administered tool used for screening, diagnosis, monitoring and measuring the severity of depression. It's composed of 9 items that correspond to the symptoms of major depression according to DSM-IV. The score has a range between 0 and 27. Scores between 0 and 9 indicate the presence of a sub-threshold depression. The score of 10 is indicated as the point at which the sensitivity and specificity of the instrument are recognized as optimal for highlighting depressions of clinical relevance.
Bodily and emotional perception of pain (BEEP), change is being assessed | T0 (0 weeks); T1 (10 weeks); T2 (22 weeks); T3 (34 weeks)
  Instrument consisting of 23 items with Likert scale with six-step interval (from 0 to 5), organized in three subscales definable according to the following denomination: Emotional reaction induced by pain (including 15 items); Limitations caused by pain in the daily life (including 4 items); and Interference of pain on mood, interpersonal relationships, sleep and pleasure of living (4 items).
Sense of Coherence Scale 13- item (SOC), change is being assessed | T0 (0 weeks); T1 (10 weeks); T2 (22 weeks); T3 (34 weeks)
  Self-administered questionnaire consisting of 13 items providing a total score and a score for each dimension: "comprehensibility" (C), which refers to the ability to perceive life events as coherent, structured and clear; "Manageability" (Ma), which refers to the ability to perceive that the available resources satisfy the needs of life; and "Significance" (Me), which refers to the feeling that life, emotionally, makes sense. The total score ranges from 13 to 91, with higher scores indicating a higher SOC.

OTHER OUTCOMES:
Quality of life, Short Form Health Survey (SF-12), change is being assessed | T0 (0 weeks); T1 (10 weeks); T2 (22 weeks); T3 (34 weeks)
  The Short Form Health Survey (SF-12), brief version of SF-36 questionnaire, made up of twelve questions, includes the following dimensions: physical activity, disturbance in physical health, physical condition, self-assessment of health status, vitality, social activity and mental health. Higher SF-12 scores recorded a greeting and QoL performance.

CONTACTS AND LOCATIONS:
Locations (1):
- P.O. San Giovanni di Dio, AOU Cagliari, Cagliari, Italy

REFERENCES:
- [Derived] Carta MG, Cossu G, Primavera D, Aviles Gonzalez CI, Testa G, Stocchino S, Finco G, Littera MT, Deidda MC, Lorrai S, Madeddu C, Nardi AE, Sancassiani F. Heart Rate Variability Biofeedback Efficacy on Fatigue and Energy Levels in Fibromyalgia: A Secondary Analysis of RCT NCT0412183. J Clin Med. 2024 Jul 9;13(14):4008. doi: 10.3390/jcm13144008. PMID 39064048
- [Derived] Carta MG, Testa G, Stocchino S, Finco G, Sancassiani F, Littera MT, Deidda MC, Ventriglio A, Bhugra D, Cossu G. The efficacy of heart rate variability biofeedback training on sleep disorders and impact of fibromyalgia: Results of a phase II randomized controlled trial. J Psychosom Res. 2024 Jun;181:111664. doi: 10.1016/j.jpsychores.2024.111664. Epub 2024 Apr 6. PMID 38652978